CLINICAL TRIAL: NCT04928430
Title: An International, Placebo-controlled, Double-blind, Randomized Clinical Trial to Evaluate the Efficacy and Safety of 150 mg XAV-19 Infusion, in Patients With Moderate to Severe COVID-19: the EUROXAV Study
Brief Title: Efficacy and Safety of XAV-19 for the Treatment of Moderate-to-severe COVID-19
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Xenothera SAS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XT-2002; 2020-005979-12 (EudraCT Number)
Record Dates: First submitted 2021-05-27; First posted 2021-06-16 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
Keywords: COVID-19; SARS-CoV-2; polyclonal IgG
MeSH Terms: conditions — COVID-19 | interventions — XAV-19

STUDY DESIGN:
Intervention Model Description: This is a phase II/III, multicenter, international, randomized (1:1), placebo-controlled, parallel group, double-blind study to evaluate the efficacy and safety of XAV-19 in patients with moderate-to-severe COVID-19.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XAV-19 (Experimental): XAV-19
  Interventions: Drug: XAV-19
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XAV-19 — 150 mg of XAV-19 single IV perfusion
  Arms: XAV-19
Drug: Placebo — Single IV infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of XAV-19 drug in patients with moderate-to-severe COVID-19.

ELIGIBILITY:
Inclusion Criteria:

I1) Male or female patient aged 18 years or over, weighing >50 Kg and <120 Kg, at the time of signing the informed consent,

I2) Patient presenting in a specialized or an emergency unit

I3) Patient presenting signs of pneumonia evidenced by at least 1 of the following: auscultation, chest X-Ray, CT scan OR presenting COVID-19 related symptoms having started less than 10 days prior to screening visit, including at least 2 of the following: fever, cough, sore throat or nasal discharge, dyspnea (shortness of breath), thoracic pain, headache or fatigue, myalgia, anosmia, dysgeusia, diarrhea, nausea

I4) Patient with SpO2 > 90% (at ambient air)

I5) Patient with a first positive SARS-CoV-2 test (RT-PCR, RT-qPCR or antigen test) in the last 10 days or at screening

I6) Women of childbearing potential (WOCBP) must have a negative urine pregnancy test at screening and use a highly effective birth control until 90 days after the administration of study drug

I7) Non-vasectomized male patients having a female partner of childbearing potential must agree to use a highly effective method of contraception until 90 days after the administration of study drug,

I8) Patient capable of giving signed informed consent.

Exclusion Criteria:

E1) Patient with a positive SARS CoV-2 test (RT-PCR, RT-qPCR or antigen test) of more than 10 days before the screening visit

E2) Patient with multiorgan failure

E3) Patient requiring immediate Intensive Care Unit (ICU) hospitalization

E4) Patient participating in another clinical trial with an investigative agent

E5) Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with an aggravation of COVID-19 | within 8 days after treatment
  The aggravation is defined as a worsening of the score of at least 1 point on the WHO 7-point ordinal scale compared to the score on the WHO 7-point ordinal scale at randomization.

SECONDARY OUTCOMES:
Change in Clinical parameters : body temperature | Between randomization and Day 3, 5, 8 and 15
  °C
Change in Clinical parameters : Respiratory rate | Between randomization and Day 3, 5, 8 and 15
  breath/min
Change in Clinical parameters : SpO2 at ambiant air | Between randomization and Day 3, 5, 8 and 15
Change in Clinical parameters : Supplemental O2 | Between randomization and Day 3, 5, 8 and 15
  L/min
Change in severity on Common Terminology Criteria of Adverse Events (CTCAE) scale (version 5.0) | Between randomization and Day 3, 5, 8 and 15
  Shortness of breath and thoracic pain
  Scale score :
  Dyspnea: grade 1 (shortness of breath with moderate exertion) to 5 (death) Non-cardiac chest pain: grade 1 (mild pain) to 3 (severe pain)
Duration of patient's requirement in supplemental O2 | up to 15 days
  Time requiring supplemental O2 at Day 15 will be defined as the time in days from randomization to the date of requiring supplemental O2.
Duration of aggravation | up to 15 days
  Duration of aggravation will be defined as the time in days between start date of aggravation and improvement date.
Length of hospital stay | up to 15 days
Viral status: RT-PCR or RT-qPCR for SARS-CoV-2 | At randomization and on Day 8 or at the end of follow-up, whichever comes first
  (positive/negative)
Proportion of patients referred to Intensive Care Unit (ICU) | Between randomization and Day 3, 5, 8 and 15
Proportion of patients with need for mechanical ventilation | At randomization and at Day 3, 5, 8 and 15
Survival rates | at day 8 and day 15 after randomization
Safety: Occurrence of adverse effects | up to 15 days
  Number and Proportion of participants with AE, SAE and treatment emergent adverse events leading to study drug discontinuation, to concomitant or additional treatment
Safety: hypersensitivity or allergy | up to 15 days
  Incidence of hypersensitivity reactions and allergy
Safety: laboratories abnormalities : white blood cell count | up to 15 days
  G/L
Safety: laboratories abnormalities : red blood cell count | up to 15 days
  10 12/L
Safety: laboratories abnormalities : hemoglobin | up to 15 days
  g/dL
Safety: laboratories abnormalities : platelets | up to 15 days
  G/L
Safety: laboratories abnormalities : creatinine | up to 15 days
  µmol/L

CONTACTS AND LOCATIONS:
Locations (18):
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment " St. Ekaterina" - Dimitrovgrad - EOOD, COVID Departement, Dimitrovgrad
  - University Multiprofile Hospital for Active Treatment - Plovdiv - AD, COVID Departement, Plovdiv
  - Complex Oncological Center - Ruse Ltd, COVID Departement, Rousse
  - Specialized Hospital for Active Treatment for Pneumophtisiatrics Diseases Dr. Dimitar Gramatikov - Ruse - EOOD, Departement of Pneumology, Rousse
  - 5th Multiprofile hospital for Active Treatment - Sofia - EAD, Departement of Pneumology and Phtisiatric, Sofia
- Greece (5):
  - Evangelismos General Hospital of Athens, Critical Care Departement, Athens
  - "Sotiria" General Hospital of Chest Diseases of Athens, 3rd Department of Medicine of University of Athens, Athens
  - University Hospital of Heraklion, Department of Internal Medicine & Infectious Diseases Unit, Heraklion
  - AHEPA University General Hospital of Thessaloniki, Infectious Diseases Division of 1st Internal Medicine Department, Thessaloniki
  - "Hippokration" General Hospital of Thessaloniki, 3rd Department of Pediatrics, Thessaloniki
- Romania (4):
  - Leon Daniello Clinical Hospital of Pneumoftiziology, Cluj-Napoca
  - Hospital for Infectious Diseases and Pneumology "Victor Babeş" Craiova, Craiova
  - Military Field Hospital ROL-2, Otopeni
  - Pius Brinzeu County Emergency Clinical Hospital Timisoara, Timișoara
- Spain (2):
  - Ramón y Cajal University Hospital, Madrid
  - Puerta del Hierro University Hospital, Majadahonda
- Turkey (Türkiye) (2):
  - Bağcılar Medipol Mega Universite Hastanesi, Bağcılar
  - Istanbul University Cerrahpasa-Cerrahpasa Medical Faculty, Fatih

REFERENCES:
- [Derived] Poulakou G, Royer PJ, Evgeniev N, Evanno G, Shneiker F, Marcelin AG, Vanhove B, Duvaux O, Marot S, Calvez V. Anti-SARS-CoV-2 glyco-humanized polyclonal antibody XAV-19: phase II/III randomized placebo-controlled trial shows acceleration to recovery for mild to moderate patients with COVID-19. Front Immunol. 2024 Apr 17;15:1330178. doi: 10.3389/fimmu.2024.1330178. eCollection 2024. PMID 38694503